CLINICAL TRIAL: NCT05558345
Title: Expression of Stress Markers in MSM Living With HIV Receiving Contingency Management for Methamphetamine Use Disorder
Brief Title: Expression of Stress Markers During Meth Treatment (EXPRESS+)
Acronym: EXPRESS+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael J. Li, PhD, MPH, Assistant Professor In-Residence, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-001564; K01DA051329 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Substance-Related Disorders; HIV
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management for Methamphetamine Reduction (Experimental): 8 weeks of contingency management, twice weekly visits, with escalating rewards from $10 to $40 for negative urine tests
  Interventions: Behavioral: Contingency Management
- Non-substance-using Control (No Intervention): Observational visits (no intervention) at baseline, Week 4, Week 8, and Week 12 for those who do not use methamphetamine.

INTERVENTIONS:
Behavioral: Contingency Management — A positive reinforcement behavioral treatment with escalating rewards for consecutive negative urine tests, starting at $10 and capped at a maximum of $40 per negative result.
  Arms: Contingency Management for Methamphetamine Reduction

SUMMARY:
This is a non-randomized behavioral trial that aims to investigate whether changes in inflammatory and type I IFN expression coincide with changes in methamphetamine use and viral load over the course of 12 weeks in HIV-positive people assigned male at birth with and without methamphetamine use disorder.

DETAILED DESCRIPTION:
This is a within-subjects, two-arm study with 35 HIV-positive people assigned male at birth receiving contingency management for treatment of methamphetamine use disorder and 20 HIV-positive people assigned male at birth serving as a non-substance-using healthy control (N=55 total). HIV-positive participants with methamphetamine use disorder who meet the eligibility criteria will be assigned to the contingency management treatment group. HIV-positive participants who do not use substances and meet the specific criteria will be assigned to the non-substance-using control group. Participants will be observed over 8 weeks, with another follow-up 4 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

For Contingency Management:

1. Assigned male sex at birth
2. 18 to 45 years of age
3. Reports having sex with men in the past 12 months.
4. HIV-positive (confirmed by certification or by HIV rapid test)
5. Has an HIV care provider (last seen in the past 12 months)
6. Has a current antiretroviral prescription
7. Meets the DSM-5 criteria for methamphetamine use disorder using SCID-5
8. Urine test is positive for methamphetamine within 30 days of their screening visit
9. Seeking treatment for methamphetamine use disorder.
10. Ability to attend twice weekly appointments for drug testing and treatment

For Non-substance-using Control:

1. Assigned male sex at birth
2. 18 to 45 years of age
3. Reports having sex with men in the past 12 months.
4. HIV-positive (confirmed by certification or by HIV rapid test)
5. Has an HIV care provider (last seen in the past 12 months)
6. Has a current antiretroviral prescription

Exclusion Criteria:

For Contingency Management:

1. Identifies as (cis- or transgender) female
2. Reports another current or past substance use disorder
3. Reports being in another intervention or clinical trial for substance use
4. Positive test for opioids, cocaine, and/or MDMA

For Non-substance-using Control:

1. Identifies as (cis- or transgender) female
2. Positive test for methamphetamine, opioids, cocaine, and/or MDMA.
3. Reports substance use (methamphetamine, opioids, cocaine, MDMA, hallucinogens, heavy alcohol use, and/or tobacco) in the past 6 months
4. Reports past or current substance use disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned male sex at birth but does not identify as female.
Enrollment: 55 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory and Type I IFN Gene Expression over 12 weeks | every 4 weeks, at baseline, Week 4, Week 8, and Week 12
  Change in gene expression values -- based on count per million or reference gene normalized mRNA extracted from leukocytes and mapped to 53 a priori specified genes -- averaged over 4 times points using mixed linear regression
Change in Methamphetamine Use over 12 weeks | twice weekly for 8 weeks with 4-week follow-up in the contingency management group; once every 4 weeks over 12 weeks for the control group.
  Change in odds of methamphetamine use -- based on qualitative urine test result -- over 12 weeks.

SECONDARY OUTCOMES:
Change in HIV Viral Suppression over 12 weeks | Once every 4 weeks over 12 weeks (i.e., baseline, Week 4, Week 8, Week 12)
  Change in odds of viral suppression -- based on viral load cut-off of < 200 c/mL blood -- over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Li, PhD, Principal Investigator — UCLA Department of Family Medicine
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
It is possible that future collaborators of the PI (e.g., other UCLA investigators) may conduct secondary analyses on the data to answer other research questions. The other investigator may submit a concept for a research question and hypothesis to be tested using the data. This would require PI approval of a concept, and co-authorship/involvement of the PI on the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the PI completes publication of their specific aims and any secondary outcomes, data will be available for at least 3 years thereafter.
Access Criteria: Submission and PI approval of a concept sheet

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT05558345/Prot_SAP_ICF_000.pdf